CLINICAL TRIAL: NCT03317587
Title: Inspiring Nutritious Selections and Positive Intentions Regarding Eating and Exercise (INSPIRE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HM20011075
Record Dates: First submitted 2017-09-27; First posted 2017-10-23 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Obesity; Eating Disorder
MeSH Terms: conditions — Obesity; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- INSPIRE (Experimental)
  Interventions: Behavioral: INSPIRE

INTERVENTIONS:
Behavioral: INSPIRE — Eight week program of weekly group sessions with homework assignments addressing beauty ideals, establishing a healthy relationship with food and exercise, and tolerating and managing uncomfortable emotions. Participants will complete questionnaires are separate time points (one week before the program, one week after the program, and 1 month after the program) to evaluate the impact of the program on various behavioral and psychological outcomes.

SUMMARY:
The aims of the current study are: 1) to pilot a manualized intervention (INSPIRE - Inspiring Nutritious Selections and Positive Intentions Regarding Eating and Exercise) to determine feasibility and acceptability, and 2) to evaluate the preliminary effectiveness of INSPIRE on physical and psychological variables.

DETAILED DESCRIPTION:
The purpose of the current study is to implement an evidence-based prevention program to promote positive health behaviors among young adult women. It will be one of the first to intentionally execute a prevention program targeting well-established risk factors for both obesity and eating disorders in this high-risk population. Intervention content focuses on promoting body size diversity and emphasizing positive health and behavior change in order to reduce stigmatization and remain sensitive to weight-related issues. The manual was developed by integrating two successful existing prevention programs and expanding on previous prevention efforts. Specifically, the diversity of beauty ideals were highlighted to enhance relevance among ethnic minority women, and distress tolerance and emotion regulation skills training were included to target the maladaptive coping mechanisms young adults use to manage the stress associated with transitioning to college.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in postsecondary education at Virginia Commonwealth University

Exclusion Criteria:

* BMI ≥ 30 kg/m2
* Meet criteria for eating disorder threshold risk
* Pregnancy

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2017-12-08 (Actual); Study Completion 2017-12-08 (Actual)

PRIMARY OUTCOMES:
Acceptability of intervention | 8 weeks
  Acceptability of the intervention will be assessed via aggregation of the ordinal-level items on the weekly participation satisfaction surveys.
Feasibility of the intervention | 8 weeks
  Feasibility of the intervention will be assessed via aggregation of the ordinal-level items on the weekly therapist feasibility surveys.

SECONDARY OUTCOMES:
Eating disorder behaviors | Baseline to 14 weeks
  Change in disordered eating behaviors will be assessed with the Eating Disorder Examination Questionnaire. Participants will complete this one week before the program, one week after the program, and one month after the program.
Risk for obesity (BMI) | Baseline to 14 weeks
  Weight will be measured (by trained staff) to the nearest ¼ kg using a digital scale and height will be measured to the nearest cm using a stadiometer; these measurements will be used to calculate BMI (kg/m2). Measurements will be taken one week before the program, one week after the program, and one month after the program.
Appearance Ideals | Baseline to14 weeks
  Changes in appearance ideals will be evaluated with the Body Image-Ideals Questionnaire, a self-report questionnaire that quantifies an individual's perceived discrepancy from and importance of internalized ideals for multiple physical attributes. Participants will complete this one week before the program, one week after the program, and one month after the program.
Emotion Regulation Difficulties | Baseline to14 weeks
  Changes in difficulty regulating emotions and tolerating distress will be assessed with the Difficulties in Emotion Regulation Scale. Participants will complete this one week before the program, one week after the program, and one month after the program.
Healthy Eating | Baseline to14 weeks
  Change in dietary intake will be assessed using the Block Food Screener, a self-report questionnaire that surveys the leading sources of fat, fiber, fruits, and vegetables in the diets of North Americans. Participants will complete this one week before the program, one week after the program, and one month after the program.
Physical Activity | Baseline to14 weeks
  Change in physical activity during the past seven days will be assessed with the Seven-Day Physical Activity Recall. This measures the frequency and duration of each physical activity performed throughout the day. Participants will complete this one week before the program, one week after the program, and one month after the program.
Thin-ideal internalization | Baseline to14 weeks
  Change in thin-ideal internalization will be assessed with the Ideal-Body Stereotype Scale - Revised. Participants will complete this one week before the program, one week after the program, and one month after the program.
Negative Affect | Baseline to14 weeks
  Change in negative affect will be assessed using the sadness, guilt, hostility, and fear/anxiety subscales of the Positive and Negative Affect Scale - Revised. Participants will complete the this one week before the program, one week after the program, and one month after the program.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Mazzeo, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Derived] Simpson CC, Burnette CB, Mazzeo SE. Integrating eating disorder and weight gain prevention: a pilot and feasibility trial of INSPIRE. Eat Weight Disord. 2020 Jun;25(3):761-775. doi: 10.1007/s40519-019-00685-w. Epub 2019 Apr 15. PMID 30982943